CLINICAL TRIAL: NCT03835520
Title: Prospective Collection of Tumor Biopsy and Plasma Samples From Cancer Patients Treated With Molecular Targeted Therapies or Immunotherapy
Acronym: Plasma-Target
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 2018-02; 2018/11JUI/248 (Registry Identifier: Ethics Committee Approval); B403201836842 (Other: Belgium Registration number)
Record Dates: First submitted 2018-10-08; First posted 2019-02-08 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Immunotherapy; Molecular Targeted Therapies; Tumor Biopsy; Plasma Samples
MeSH Terms: conditions — Neoplasms | interventions — Adjuvants, Immunologic; Rv1579c phage protein, Mycobacterium tuberculosis

STUDY DESIGN:
Intervention Model Description: The trial will include patients with any type of cancer treated with one of the following regimens after signing of the patient's informed consent:
  * I: Molecular targeted agent
  * II: Immunotherapy
Masking Description: Masking and allocation tbc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOLECULAR TARGETED THERAPIES (Experimental): Immunotherapy will be administered according to standard of care and reimbursement modalities in Belgium. Targeted agents will be administered according to manufacturer's instructions.
  Interventions: Drug: Molecular Target
- IMMUNOTHERAPY (Experimental): Immunotherapy will be administered according to standard of care and reimbursement modalities in Belgium.
  Interventions: Drug: Immunotherapeutic Agent

INTERVENTIONS:
Drug: Immunotherapeutic Agent — Immunotherapy will be administered according to standard of care and reimbursement modalities in Belgium.
  Arms: IMMUNOTHERAPY
Drug: Molecular Target — Targeted agents will be administered according to standard of care and reimbursement modalities in Belgium. Targeted agents will be administered according to manufacturer's instructions.
  Arms: MOLECULAR TARGETED THERAPIES

SUMMARY:
The purpose of this study is to collect blood samples, as well as tumor tissue for genetic analysis. The collection of samples will allow the creation of a plasma bank. Targeted individuals are cancer patients of all types, treated with immunotherapy or targeted therapy.

Immunotherapy or targeted agents will be administered according to standard of care and reimbursement modalities in Belgium. Targeted agents will be administered according to manufacturer's instructions.

With the aim to identify predictive markers of response to treatment or possible resistance mechanism, the plasma samples and the tumor samples will be used for genetic analysis, for example but not limited to, whole exome sequencing. This may lead to the discovery of some germinal mutations implicated in other diseases than cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer treated with one of the following regimens: Molecular targeted agents or Immunotherapy
* Paraffin-embedded tumor tissue available for immunohistochemistry and/or DNA extraction.
* Patient able to give written informed consent.

Exclusion Criteria:

* Patients with cancer treated with other regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of treatment against Cancer | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Efficacy will be determined in terms of overall responses according to standard practice by the local investigator. Disease and response assessments are defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of first documented progression assessed up to 120 months
  Overall survival is defined as the time from the date of inclusion to the date of death from any cause or to the date of last follow-up (in exceptional cases where it is impossible to document the date of death). Every effort should be made to document the cause of death.
Progression free survival | From date of randomization until the date of first documented progression , assessed up to 120 months
  Progression free survival (PFS) will be measured from the date of inclusion to the date of progression or death, whatever the cause.
  Progression will be defined according to the RECIST criteria.
Objective tumor response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Objective tumor response will be measured according to the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No